CLINICAL TRIAL: NCT01753765
Title: A Prospective Non-Randomized Unblinded Study Evaluating the Treatment of Occipital Neuralgia With the Cryo-Touch III Device
Brief Title: Study Evaluating the Treatment of Occipital Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYO-0613
Record Dates: First submitted 2012-12-14; First posted 2012-12-20 (Estimated); Results first posted 2023-06-05 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Occipital Neuralgia
Keywords: occipital neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Study treatment with Cryo-Touch III device at Day 0.
  Interventions: Device: Device: Cryo-Touch III Study treatment at Day 0.

INTERVENTIONS:
Device: Device: Cryo-Touch III Study treatment at Day 0. — Device: Cryo-Touch III Study treatment at Day 0.

SUMMARY:
A proof of concept study to evaluate the feasibility of safe and effective treatment through optimization of the Cryo-Touch III device for temporary relief of or reduction in pain due to occipital neuralgia.

DETAILED DESCRIPTION:
Over 100 million patients in the United States suffer from chronic pain. Chronic pain conditions are often debilitating, taking a toll on a patient's physical and mental welfare. Though a variety of pain management techniques currently exist, the most common nonsurgical options provide slow-acting and/or short-term relief. Medication, often in the form of non-steroidal anti-inflammatory drugs (NSAIDs) and opioids, comes with an array of side effects such as nausea and vomiting. Medication also presents the possibility of more serious effects such as increased risk of heart attack and stroke, and tolerance or dependency issues. Surgical strategies tend to be reserved for more severe cases and are limited by the risks and complications typically associated with surgery including bleeding, bruising, scarring, and infection. A nonsurgical, minimally invasive, long-lasting approach to chronic pain management is desirable.

Myoscience, Inc. (Redwood City, CA) has developed a pain management device - the Cryo-Touch III - for a novel, minimally invasive procedure using focused cold therapy to target sensory nerve tissue and offer long-lasting pain relief through cryoanalgesia. The device operates on the well-established cryobiology principle that localized exposure to controlled, moderately low temperature conditions can alter tissue function. The therapy treats nerves via a probe in the form of an assembly of small diameter needles, creating a highly localized, low temperature treatment zone around the probe. This focused cold therapy creates a conduction block that prevents nerve signaling. Prior studies of the Cryo-Touch, Cryo-Touch II, Cryo-Touch III (a.k.a. PCP 1.0) devices have provided preliminary evidence of effectiveness on motor nerves and have been shown to be safe with no serious device-related adverse events.

Though studies have proven efficacious in targeting motor nerves, the device's effect on sensory nerves has yet to be investigated in the clinical setting. The goal of the study described herein is to evaluate the degree and duration of effect of the Cryo-Touch III in reducing chronic pain by targeting sensory nerves.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age and older. Female subjects of childbearing potential must not be pregnant at time of treatment.
2. A confirmed diagnosis of occipital neuralgia (unilateral or bilateral) .
3. Any medication must be maintained on a stable schedule for at least two weeks prior to treatment. No washout period is allowed.
4. Must have an average score for pain of ≥ 4/10 Visual Analog Scale (VAS) over the last 7 days.
5. Subject is willing and able to give written informed consent and able to comply with study instructions.

Exclusion Criteria:

1. Current diagnosis of fibromyalgia, chronic back pain, or chronic migraines.
2. Any injections intended for pain relief or neuromodulation to the upper trunk or head within the last 3 months.
3. History of a cerebrovascular accident (CVA), head trauma, stroke, or bone deformity.
4. Patient who has severe pain for any reason other than occipital neuralgia.
5. Any use of (i.e. oral, topical, inhaled and/or injected) anesthetics or steroids within the last 30 days.
6. Any previous surgery in the intended treatment area.
7. Currently enrolled in any other investigational drug or device study or participation within the last 30 days.
8. Any clotting disorder and/or use of any anticoagulant (e.g., warfarin, clopidogrel, etc.) within seven (7) days prior to administration of the treatment.
9. Allergy or intolerance to any preparatory treatment agent or any other substance utilized within the study.
10. Any local skin condition at the treatment site that would adversely affect treatment or subject safety.
11. Any confounding diagnosis or medical condition that in the investigator's opinion would adversely affect study participation or subject safety.
12. Any chronic medication use (prescription, over-the-counter, supplements, etc.) that in the investigator's opinion would adversely affect study participation or subject safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Neurovations, Napa, California
  - Injury Care Medical Center, Boise, Idaho
  - International Clinical Research, Overland Park, Kansas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 26
Average baseline Pain Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — VAS Scoring is 0-10 where 0 equals no pain and 10 is the highest score possible. Higher scores equate to worse outcome.
  units on a scale | 6.3 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: A Reduction in Either Pain Frequency or Severity Associated With Occipital Neuralgia.
Description: Improvement of pain due to occipital neuralgia as measured on the Visual Analog Scale (VAS) for pain at Days 7 and 30 as compared to baseline (Day 0). 0= no pain, 10= worst pain imaginable. Higher scores equal worse outcome.
Time Frame: Baseline to Day 7, Baseline to Day 30
Population: The variation in number analyzed at each timepoint from overall number of patients analyzed is due to the reflection of the actual number of participants with data collected at specified timepoint.
Measure: Mean (Standard Deviation); unit: point improvement
Arm/Group | Treatment
Number analyzed (Participants) | 26
point improvement
  Average Point Improvement Day 7: number analyzed (Participants) | 25
  Average Point Improvement Day 7 | 2.5 (2.5)
  Average Point Improvement Day 30: number analyzed (Participants) | 23
  Average Point Improvement Day 30 | 2.7 (2.2)

2. Secondary Outcome: Duration of Treatment
Description: Treatment effect was based on Subject response when asked if the Subject had an effect from the treatment.
Time Frame: Day 30, Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 26
Participants
  Day 30 | 13
  Day 56 | 9

ADVERSE EVENTS:
Time Frame: Adverse events will be recorded from initiation of study treatment to Visit 5 Day 56- end of study
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 5/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=26)
Cold (Infections and infestations) | 1 (1)
Dizziness secondary to oral gabapentin medicine (General disorders) | 1 (1)
Increased knee pain secondary to fall (Injury, poisoning and procedural complications) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 1 (1)
pain in treatment area (Injury, poisoning and procedural complications) | 1 (1)
increased pain in neck area (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less